CLINICAL TRIAL: NCT02451462
Title: Trial of Zoledronic Acid to Prevent Bone Loss in Hematopoietic Cell Transplant Recipients
Brief Title: Pilot Trial of Zoledronic Acid to Prevent Bone Loss in Hematopoietic Cell Transplant Recipients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VAR0122-BMT290; 31259
Record Dates: First submitted 2015-05-15; First posted 2015-05-22 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Hematopoietic Stem Cell Transplant; Bone Marrow Transplant
Keywords: hematopoietic stem cell transplant; bone marrow transplant
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zoledronic acid arm (Experimental): Zoledronic acid
  Interventions: Drug: Zoledronic acid
- placebo arm (No Intervention): placebo

INTERVENTIONS:
Drug: Zoledronic acid
  Arms: Zoledronic acid arm

SUMMARY:
Patients who undergo bone marrow transplant for different types of cancer are exposed to many treatments such as steroids and whole body radiation. These treatments make the transplant possible but also make their bones weaker and more prone to fractures which can be a source of significant disability and decreased quality of life for cancer survivors. Our trial will investigate whether giving one dose of Zoledronic acid (a commonly used drug given to preserve bone mass in osteoporosis) before bone marrow transplant can protect from the bone loss caused by the transplant procedures. The investigators are also interested in studying the complex interactions of bone, muscle and fat which are greatly affected after bone marrow transplant.

DETAILED DESCRIPTION:
Primary Objective:

To determine whether a single dose of zoledronic acid pre-transplant will prevent HSCT-related bone loss without impeding engraftment, compared with placebo.

Secondary Objectives:

To identify bone and muscle deficits and alterations in fat distribution prior to HSCT, compared with healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* First allogeneic HSCT
* Age > 18 years
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Current or prior use of bone active medication (bisphosphonates, teriparatide, selective estrogen receptor modulators, or Denosumab)
* Hypo- (Ca < 8.5 mg/dL) or hyper-calcemia (Ca > 10.5 mg/dL)
* Hyperthyroidism (TSH < 0.4 mIU/L and free T4 > 1.6 ng/dL)
* Hyperparathyroidism (PTH > 80 pg/mL)
* Estimated GFR < 35 ml/min/1.73 m2
* Other chronic disease unrelated to HSCT that may impact bone metabolism
* Osteoporosis: patients with a history of fragility fracture, or a Hip or Spine T score of <-2.5 (these patients will be treated with Zoledronic Acid and followed, but excluded from randomization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
% change in Bone Mineral Density at the Femoral Neck | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Joy Wu, Principal Investigator — Stanford University